CLINICAL TRIAL: NCT03691688
Title: The Long Term Effect of Low Dose Aspirin on Uric Acid in Chinese Patients With Coronary Artery Disease（AURORA): A Prospective Cohort Study
Brief Title: The Long Term Effect of Low Dose Aspirin on Uric Acid in Chinese Patients With Coronary Artery Disease（AURORA）
Acronym: AURORA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Chief of Cardiology Department, Shanghai Zhongshan Hospital
Other Study IDs: ZS-AURORA
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease; Hyperuricemia
Keywords: aspirin; coronary artery disease, uric acid
MeSH Terms: conditions — Coronary Artery Disease; Hyperuricemia | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspirin: Aspirin 100mg
  Interventions: Drug: Aspirin 100 mg
- Clopidogrel: Clopidogrel 75mg
  Interventions: Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Aspirin 100 mg — Aspirin 100mg will be prescribed for antiplatelet therapy at the physician's discretion
  Groups: Aspirin
Drug: Clopidogrel 75mg — Clopidogrel will be prescribed for antiplatelet therapy in case of aspirin intolerance at the physician's discretion
  Groups: Clopidogrel

SUMMARY:
The deleterious effects of hyperuricemia (HUA) on cardiovascular disease (CVD) were well established. Aspirin is the most commonly prescribed antiplatelet agent for primary or secondary prophylaxis of CVD. Only a few short-term studies in the elderly suggested low-dose aspirin, e.g., 75-100 mg/day, increases serum urate by reducing urinary uric acid excretion. However, monitoring of renal function is currently not recommended. Little is known about the long-term effect of low dose aspirin on uric acid. The principal aim of this prospective cohort study therefore is to evaluate the renal effects of long-term aspirin (100 mg/d) administration in Chinese patients with coronary artery disease or other CVDs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with coronary artery disease (CAD) who underwent (Percutaneous Transluminal Coronary Intervention) PCI therapy, documenting angiographically at least one vessel stenosis ≥50% among major coronary arteries (left main, left anterior descending, left circumflex or right coronary artery) , manifesting clinically as latent CAD, stable CAD, unstable CAD, and acute myocardial infarction.
2. Patients with CAD without PCI therapy. They document angiographically at least one vessel stenosis ≥50% among major coronary arteries (left main, left anterior descending, left circumflex or right coronary artery) , and classified clinically as latent CAD, stable CAD, unstable CAD.
3. Patients without CAD who needs antiplatelet therapy for prophylaxis of ASCVD, documenting angiographically no vessel stenosis ≥50% among any of major coronary arteries (left main, left anterior descending, left circumflex or right coronary artery).

Exclusion Criteria:

1. Patients with severe conditions with life expectancy less than 12 months.
2. Patients with malignant tumor.
3. Severe Kidney disease: patients with acute kidney injury, nephritic syndrome, renal replacement therapy, kidney transplant or eGFR <30 mL/min/1.73 m2.
4. Contraindicated to antiplatelet therapy because of acute bleeding.
5. Patients who formerly administrated aspirin for at least one week or withdrawal of aspirin less than one month before enrollment.
6. Patients who formerly administrated UA lowering agents at least one month before enrollment.
7. Patients who formerly administrated, stopped or titrated doses of any of the following drugs at least one month before enrollment: losartan, irbesartan, fenofibrate, thiazide and loop diuretics.
8. Patients who administrated ticagrelor as antiplatelet agent one month before enrollment or since then.

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of angiographically diagnosised CAD patients with or without PCI, and patients without CAD who needs antiplatlet therapy for prophylaxis of ASCVD.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
HUA ( serum uric acid level, μmol/L) | 24 months after enrollment
  Two different days of fasting uric acid >420 μmol/L and women >360 μmol/L under normal purine diet.
Gout attacks (ACR/EULAR classification criteria 2015) | 24 months after enrollment
  Gout attacks are confirmed according to ACR/EULAR classification criteria 2015
Initiation of UA-lowering agents | 24 months after enrollment
  Starting febuxostat, allopurinol,or benzbromarone therapy at physicians' descretion

SECONDARY OUTCOMES:
Renal impairment (serum creatine level, μmol/L) | 24 months after enrollment
  2-fold elevation of serum creatine level from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, Study Chair — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No